CLINICAL TRIAL: NCT02717845
Title: Computerized Tomography (CT) Scan Study of Bone Healing Following Open Wedge Proximal Tibial Osteotomy [CT Imaging Study for Knee Osteotomy (CISKO)]
Brief Title: CT Imaging Study for Knee Osteotomy (CISKO)
Acronym: CISKO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: North Cumbria University Hospitals NHS Trust (Other)
Collaborators: NuVasive (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PR0251; 16/NW/0038 (Other: UK National Research Ethics Service)
Record Dates: First submitted 2016-03-15; First posted 2016-03-24 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Bone Malalignment
Keywords: varus malignment; osteoarthritis; knee
MeSH Terms: conditions — Bone Malalignment; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CT scan Ellipse (Experimental): New medical device for high tibial osteotomy
  Interventions: Device: Ellipse
- CT scan Tomofix (Active Comparator): Established medical device for high tibial osteotomy
  Interventions: Device: Tomofix

INTERVENTIONS:
Device: Ellipse — diagnostic CT scan imaging
  Arms: CT scan Ellipse
Device: Tomofix — diagnostic CT scan imaging
  Arms: CT scan Tomofix

SUMMARY:
Malalignment of the knee joint causes arthritis in later life. Currently there are three surgical ways to treat knee arthritis: total knee replacement, partial knee replacement, and high tibial osteotomy (HTO). The former two very much focus on treating the effect of malalignment, i.e. removing the arthritic joint. However, HTO addresses the cause of the arthritis, namely the joint malalignment. This preserves the patient's joint and it means that a patient will start using the unaffected part of the knee joint more.

HTO involves cutting a wedge out the tibia to correct the alignment of that bone with the knee joint, to redistribute load from the affected medial part to lateral part. To keep the tibia in the new position, a medical nail device is attached to keep it in place and allow new bone to regenerate within the wedge. Currently, the market leader for HTO is the TomoFix (by DePuySynthes company) plate and nail device. As the name suggests, TomoFix is fixed at surgery and therefore the change in bone angle cannot be changed afterwards. It does mean that patients can be weight-bearing on the affected leg soon after the HTO procedure. A new CE-marked device is being tested in an interventional trial; it is produced by Ellipse Technologies. This device is an extendable nail and inserted intramedullary; following surgery the nail is tend slowly extended over a period of time until the bone correction is satisfactory.

The CISKO imaging study will assess whether there is a difference between the TomoFix and Ellipse system in terms of bone regeneration in the tibial wedge by performing a CT-scan at 3 and 6 months post-operatively. This will be quantified by two independent radiological reports. A secondary objective is to investigate patient satisfaction and also patient pain levels at these time intervals. The degree of bone healing is usually the main factor holding clinicians back when it comes to advising patients on what activities they can return to post-operatively. A difference in bone healing between the two systems may impact on the advice clinicians can give patients regarding recommencing more intense activities such as recreational sports, which ultimately could positively impact patients' health and well-being.

DETAILED DESCRIPTION:
One treatment modality for medial osteoarthritis of the knee is open-wedge high tibial osteotomy (HTO). The current most common way of performing HTO is to use fixation plates with locking bolts implanted in the patient's tibia, to allow increased stability & joint movement and the ability to be weight bearing on the affected leg sooner . However, despite advances in high tibial osteotomy technology, it can still take most patients about six months to fully recover from the procedure. Sedentary activities are usually picked up about a month after surgery, before physical work is introduced 3 to 4 months after surgery, followed by sports which can be reintroduced approximately 6-12 months after surgery. One reservation for allowing patients to be fully weight bearing early on is the perceived risk of loss of correction of the angle, although in practice this effect appears to be a rare occurrence . For example, in a series of patients Takeuchi and colleagues showed that full weight-bearing is possible two weeks after surgery without implications for the correction made to the joint angle .

It is imperative that the open wedge is healed and repopulated by new bone, to strengthen the tibia and allow full recovery following HTO. Regeneration will take place naturally, although some surgeons apply aids to promote bone healing, such as the ChronOS β-tricalcium phosphate wedge. However, research into this aspect of filling the wedge has shown that there is no advantage to using the filler - both in terms of stability and bone healing time of the wedge . Although fixed systems like Tomofix facilitate early weight-bearing of the affected joint, the complete closure and consolidation of the wedge takes considerably longer. In one study, 23 /27 (85%) osteotomies were fully healed twelve months after procedure . Histologically, there is variability in the degree of healing and indeed maturation of bone regeneration achieved in the tibial wedge. With current fixed plate devices, even two years post-procedure, a minor subset of patients will not have significant signs of regeneration in the surgical site. In the majority of patients, partial bone regeneration with fibrocartilaginous tissue takes place and in some patients by new regenerated fibrocartilage or hyaline-like cartilage will appear .

HTO could be improved upon to allow an earlier return to activities by patients and to achieve better rates of healing - both in terms of time and maturity of the regenerated bone. Ellipse Technologies have devised a new nail system for high tibial osteotomy that differs from the established 'locked' plate and nail systems. Their system functions in a more gradual fashion. The wedge is created in the tibia as per normal but then the Ellipse nail is inserted and per day the nail is extended in small measures (appr 1.5 mm per day) until the desired correction has been achieved. Currently the new Ellipse system is being trialed in various countries in Europe, including the Netherlands and the UK. The main Ellipse trial is seeking to establish whether the corrective power of this medical device is more accurate than the plate/nail systems in use at present. The degree of bone regeneration in the open wedge is reported on, but not in detail - e.g. by one reporting radiologist - and by using standard X-ray imaging which is primarily used for angle measurements.

This present study seeks to explore in more detail how the Tomofix and Ellipse high-tibial osteotomy systems function in relation to bone regeneration in the open-wedge created as part of the procedure by utilising CT imaging techniques rather than standard clinical X-ray imaging. The primary aim of osteotomy is realignment of the joint and thereby preserves the joint so that the patient can continue to enjoy the active life style, sports and recreational activities. After an osteotomy procedure, whenever a patient asks for advice to the clinician when they can start participating in unrestricted sports activities, clinicians often find it very difficult to answer this question. This is primarily because it is often very difficult to quantify the bone healing process precisely on radiographs. By quantifying the amount of bone healing on CT scan which is more clear and accurate, the clinician can confidently advise the patient regarding the participation in various sports activities without ambiguity.

Further, by comparing the bone healing process between Tomofix plate and Ellipse nail, investigators can make more informed judgement regarding their performance. This research will also enhance the choice of implant selection in osteotomy patients based on the duration of bone healing.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. Males
3. Mental capacity

Exclusion Criteria:

1. Under age (< 18 years)
2. Patients lacking mental capacity.
3. Females
4. Current use of nicotine products.
5. Patients who cannot understand English and therefore cannot be consented.

Pre-existing clinical exclusion criteria (for both Ellipse and Tomofix patients):

1. Varus deformity greater than 10°
2. Flexion contracture greater than 15°
3. Knee flexion under 90°
4. Medial/lateral tibial subluxation over 1 cm
5. Medial bone loss of over 3 mm
6. Inflammatory arthritis (including use of methotrexate)
7. Arthritis in the lateral compartment
8. Patella baja
9. Weight over 114 kg
10. Severe patella femoral symptoms
11. Unaddressed ligamentous instability
12. Fixed flexion contracture
13. Known or suspected osteoporosis or osteopenia based on medical history and radiographic image
14. Requires other surgical procedures at the time of the HTO surgery -

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-01 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Healing score | 3 months
  Healing of the osteotomy site after final correction as assessed by two independent radiology reports based on visual assessment of the CT imaging

SECONDARY OUTCOMES:
Patient satisfaction score | 6 months
  Patients' perspective of the degree of healing and rehabilitation following high tibial osteotomy
Change in KOOS score | 6 months
  difference in KOOS score , comparing per-operative vs 6 months post-operative.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Hafner, PhD, Study Director — NuVasive
Locations (1):
- Cumberland Infirmary, Carlisle, Cumbria, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Results to be published in peer-reviewed scientific journal